CLINICAL TRIAL: NCT03541798
Title: Comparison of Three Different Sitting Positions for Performing Combined Spinal-Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Ceyda Ozhan Caparlar, Director, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 49/08
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural; Hip Arthropathy; Knee Arthropathy
Keywords: traditional sitting position; combine spinal-epidural anesthesia; orthopedic surgery

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional sitting position (Active Comparator): Patient is positioned with her knees flexed 90o, both feet hanging of the bed and propped up by a chair, both arms hugging a pillow, adducted pelvic, maximum pelvic flexion were done to create maximal sagittal lumbal flexion before spinal anesthesia begun.
  Intervention: A combined spinal epidural anesthesia (CSE) will be applied using a CSE Tuohy Needle (18 G) and 27 G Whitacre spinal needle via needle - through needle technique. The epidural space will be located with loss of resistance to saline. 3 ml hyperbaric bupivacaine 0.5% (15 mg) will be given for spinal anesthesia.
  Interventions: Procedure: positions of patients for combined spinal-epidural anesthesia; Procedure: Combined spinal epidural anesthesia
- Harmstring stretch position (Experimental): the patients sit up from supine position with the legs remaining on the operating table, knees are maximally extended.
  Intervention: A combined spinal epidural anesthesia (CSE) will be applied using a CSE Tuohy Needle (18 G) and 27 G Whitacre spinal needle via needle - through needle technique. The epidural space will be located with loss of resistance to saline. 3 ml hyperbaric bupivacaine 0.5% (15 mg) will be given for spinal anesthesia.
  Interventions: Procedure: positions of patients for combined spinal-epidural anesthesia; Procedure: Combined spinal epidural anesthesia
- Squatting position (Experimental): the patients sit up from supine position with the legs remaining on the operating table, hips and knees are maximally flexed .
  Intervention: A combined spinal epidural anesthesia (CSE) will be applied using a CSE Tuohy Needle (18 G) and 27 G Whitacre spinal needle via needle - through needle technique. The epidural space will be located with loss of resistance to saline. 3 ml hyperbaric bupivacaine 0.5% (15 mg) will be given for spinal anesthesia.
  Interventions: Procedure: positions of patients for combined spinal-epidural anesthesia; Procedure: Combined spinal epidural anesthesia

INTERVENTIONS:
Procedure: positions of patients for combined spinal-epidural anesthesia — Patients in groups will be positioned according to the study groups for performing combined spinal epidural anesthesia.
Procedure: Combined spinal epidural anesthesia — After positioning, a combined spinal epidural anesthesia (CSE) will be applied using a CSE Tuohy Needle (18 G) and 27 G Whitacre spinal needle via needle - through needle technique. The epidural space will be located with loss of resistance to saline. 3 ml hyperbaric bupivacaine 0.5% (15 mg) will be given for spinal anesthesia after identification of subarachnoidal space.

SUMMARY:
In this prospective and randomized study, we aimed to compare the effect of of three sitting positions (the traditional sitting position (TSP), the harmstring stretch position (HSP), and the squatting position on the success rate of combined spinal epidural anesthesia in patients undergoing total knee arhtoplasty (TKA) or total hip arthroplasty (THA) surgery.

DETAILED DESCRIPTION:
Positioning of patients plays a major role to identify accurately epidural and/or spinal spaces for neuraxial blocks. Flexed back is considered mandatory to widen the inter spinous space in traditional lateral and sitting positions. In traditional sitting position (TSP), the patient is positioned in a sitting posture on the operating table. A stool is placed by the side of the operating table to support the legs. Both hips and knees are maximally flexed.

In recent years, several studies suggested that the reduction of lumbar lordosis may increase the success rate of spinal or epidural block and reduce needle-bone contact. Different modified sitting positions were described for this aim: the harmstring stretch position (HSP), the squatting position (SP), and the crossed-leg position (CLP).

In modified sitting positions, the patients sit up from supine position with the legs remaining on the operating table, either knees are maximally extended (the harmstring stretch position), or hips and knees are maximally flexed (the squatting position), or hips and knees are flexed with crossing the legs (the crossed leg position). All studies comparing modified sitting positions with TSP found that the success rate and number of needle bone contacts were similar except one study which reported a lower needle bone contact with squatting position. Other factors contributing the success of the neuraxial block were: anatomical landmarks (palpability of the spinous processes, identification of the midline), immobilization of the patient during the injection, and the provider's level of experience.

The combined spinal - epidural (CSE) technique has been increasingly used for over thirty years which consist of intentional injection of a local anesthetic into the subarachnoidal space and the placement of a catheter into epidural space to prolong or modify the block.

Although CSE technique combines the best features of spinal and epidural blockade, it is a more complicated to perform. Studies comparing CSE with epidural and/or spinal technique reported similar failure rates but most of them did not focuse on the effect of patient's positioning.

In this prospective and randomized study, we aimed to compare the effect of of three sitting positions (the traditional sitting position (TSP), the harmstring stretch position (HSP), and the squatting position (SP) on the success rate of CSE anesthesia in patients undergoing total knee arhtoplasty (TKA) or total hip arthroplasty (THA) surgery. The CLSP was not included in the study design because the crossing the legs during the procedure seemed to be painful and difficult in patients with degenerated knee joints.

Our primary endpoint was the number of needle bone contact and the secondary endpoint was ease of needle insertion/space identification.

ELIGIBILITY:
Inclusion Criteria: ASA I-II, 18-70 years, combine spinal-epidural anesthesia for elective orthopedic surgery

Exclusion Criteria: hypertension, thrombocytopenia, high intracranial pressure, Alzheimer Disease, local anesthetic allegic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Ease of identifying of epidural and subarachnoidal space | 3 months
  After positioning of patients for CSE according to groups, the block performer will palpate the iliac crest on both sides. The horizontal line between iliac crests will be used to define the level of the lumbar vertebrae. The lumbar spinous processes of L2, L3,L4, and L5 vertebra levels will be palpated and the palpability of the spinous processes will be graded by the performer to find - out best and the second best interspinous space between spinous processes as follows: easily palpable(score=2), hardly palpable (score=1) and impalpable (score=0). An interspinous space with two easy palpable spinous process will be defined as best interspinous space.An interspinous space with one easy palpable spinous process and a hardly palpable spinous processes will be defined as second best interspinous space. When all spinous processess are impalpable, the performer should choose an interspinous space to perform CSE.

SECONDARY OUTCOMES:
The number of epidural needle-bone contact | 3 months
  The number of epidural needle-bone contact for each positions

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Ö caparlar, Study Director — Dıskapı TRH; mehmet Ozhan, Study Chair — private cankaya hospital, Ankara
Locations (1):
- University of Health Dıskapı Yıldırım Beyazıt Training and Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soltani Mohammadi S, Hassani M, Marashi SM. Comparing the squatting position and traditional sitting position for ease of spinal needle placement: a randomized clinical trial. Anesth Pain Med. 2014 Apr 5;4(2):e13969. doi: 10.5812/aapm.13969. eCollection 2014 May. PMID 24790901
- [Result] Soltani Mohammadi S, Piri M, Khajehnasiri A. Comparing Three Different Modified Sitting Positions for Ease of Spinal Needle Insertion in Patients Undergoing Spinal Anesthesia. Anesth Pain Med. 2017 Oct 23;7(5):e55932. doi: 10.5812/aapm.55932. eCollection 2017 Oct. PMID 29696117
- [Result] Fisher KS, Arnholt AT, Douglas ME, Vandiver SL, Nguyen DH. A randomized trial of the traditional sitting position versus the hamstring stretch position for labor epidural needle placement. Anesth Analg. 2009 Aug;109(2):532-4. doi: 10.1213/ane.0b013e3181ac6c79. PMID 19608828
- [Derived] Ozhan MO, Caparlar CO, Suzer MA, Eskin MB, Atik B. Comparison of three sitting positions for combined spinal - epidural anesthesia: a multicenter randomized controlled trial. Braz J Anesthesiol. 2021 Mar-Apr;71(2):129-136. doi: 10.1016/j.bjane.2020.12.012. Epub 2020 Dec 28. PMID 33894856